CLINICAL TRIAL: NCT02915783
Title: A Single-arm, Multicenter, Phase 2 Trial to Evaluate Efficacy and Safety of Lenvatinib in Combination With Everolimus in Subjects With Unresectable Advanced or Metastatic Non Clear Cell Renal Cell Carcinoma (nccRCC) Who Have Not Received Any Chemotherapy for Advanced Disease
Brief Title: A Trial to Evaluate Efficacy and Safety of Lenvatinib in Combination With Everolimus in Subjects With Unresectable Advanced or Metastatic Non Clear Cell Renal Cell Carcinoma (nccRCC) Who Have Not Received Any Chemotherapy for Advanced Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-M001-221
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2021-06

CONDITIONS: Non Clear Cell Renal Cell Carcinoma (nccRCC)
Keywords: unresectable advanced; metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — lenvatinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lenvatinib 18 mg/day and everolimus 5 mg/day (Experimental): Participants will receive initial doses of lenvatinib 18 milligrams per day (mg/day) (one 10-mg capsule and two 4-mg capsules) and everolimus 5 mg/day (5-mg tablets). Capsules and tablets are to be taken orally in immediate succession once a day (QD), and dosing is recommended to occur at approximately the same time each morning (consistently either with or without food).
  Interventions: Drug: lenvatinib; Drug: everolimus

INTERVENTIONS:
Drug: lenvatinib — 4 mg and 10 mg capsules
Drug: everolimus — 5 mg tablets

SUMMARY:
This is a single-arm, multicenter, Phase 2 study of lenvatinib in combination with everolimus in participants with unresectable advanced or metastatic non clear cell renal cell carcinoma (nccRCC) who have not received any chemotherapy for advanced disease. The primary objective of the study is to evaluate the objective response rate (ORR). This study consists of three phases: a Pretreatment Phase (Screening and Baseline Periods), a Treatment Phase (starting Cycle 1, Day 1), and a Posttreatment Phase (End of Treatment Visit and survival Follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥18 years at the time of informed consent form (ICF)
* Participants with histologically confirmed non clear cell renal cell carcinoma (nccRCC) who have not received any chemotherapy for advanced disease. Participants must have one of the following subtypes of nccRCC: papillary, chromophobe, collecting duct carcinoma (CDC), renal medullary carcinoma (RMC), or unclassified.
* Radiologically measurable disease meeting the following criteria:

  1. At least 1 lesion of ≥10 millimeters (mm) in the longest diameter for a nonlymph node or ≥15 mm in the short axis diameter for a lymph node that is serially measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 using computerized tomography (CT) or magnetic resonance imaging (MRI);
  2. Lesions that have had external beam radiotherapy (EBRT) or locoregional therapies such as radiofrequency (RF) ablation must show evidence of subsequent progressive disease (substantial size increase of ≥20%) to be deemed a target lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Blood pressure (BP) ≤140/90 millimeters of mercury (mmHg) at Screening with or without antihypertensive medications and no change in antihypertensive medications within 1 week prior to Cycle 1/Day 1.
* Adequate renal function as evidenced by calculated creatinine clearance ≥30 milliliters (mL)/minute according to the Cockcroft and Gault formula
* Adequate bone marrow function:

  1. Absolute neutrophil count (ANC) ≥1.5 × 10^9/liter (L);
  2. Hemoglobin ≥10.0 grams per deciliter (g/dL) (can be corrected by growth factor or transfusion prior to first dose of study drug);
  3. Platelet count ≥100 × 10^9/L
* Adequate liver function:

  1. Bilirubin ≤1.5 × upper limit of normal (ULN) except for unconjugated hyperbilirubinemia or Gilbert's syndrome;
  2. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3 × ULN (≤5 × ULN if participant has liver metastases). If ALP is >3 × ULN (in the absence of liver metastases) or >5 × ULN (in the presence of liver metastases) AND participants are also known to have bone metastases, the liver-specific ALP must be separated from the total and used to assess the liver function instead of the total ALP.
* Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol

Exclusion Criteria:

* Predominant clear cell renal cell carcinoma (RCC)
* Prior anticancer chemotherapy or targeted therapy for advanced nccRCC
* Prior exposure to lenvatinib or mammalian target of rapamycin (mTOR) inhibitor
* Known intolerance to lenvatinib, everolimus (or other rapamycin derivatives), or any of the excipients
* Major surgery performed within 3 weeks prior to the first dose of study drugs or scheduled for major surgery during the study
* Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib or everolimus
* Participants having >1+ proteinuria on urine dipstick testing will undergo 24 hour urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥1 grams (g)/24 hours will be ineligible.
* Fasting total cholesterol ˃300 milligrams (mg)/dL (or ˃7.75 millimoles [mmol]/L) or fasting triglycerides level ˃2.5 × ULN. Note: these participants can be included after initiation or adjustment of lipid-lowering medication.
* Uncontrolled diabetes as defined by fasting glucose >1.5 times the ULN. Note: In case this threshold is exceeded, these participants can only be included after initiation or adjustment of glucose-lowering medication.
* Known history of, or any evidence of, interstitial lung disease or active noninfectious pneumonitis.
* Significant cardiovascular impairment: history of (a) congestive heart failure greater than New York Heart Association (NYHA) Class II; (b) unstable angina; (c) myocardial infarction; (d) stroke; or (e) cardiac arrhythmia associated with hemodynamic instability within 6 months of the first dose of study drugs
* Prolongation of QTcF interval to >480 milliseconds (msec)
* Known history of human immunodeficiency virus (HIV) positive
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] RNA detected)
* Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Participants with central nervous system (CNS) (e.g., brain or leptomeningeal) metastases.
* Other active malignancy (except definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or bladder) within the past 24 months
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 International Units [IU]/L or equivalent units of β-hCG or hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Females of childbearing potential who:

  1. Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as a condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 28 days after study drug discontinuation
  2. Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from being sexually active during the study period or for 28 days after study drug discontinuation
  3. Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation
  4. Are using oral hormonal contraceptives and who do not agree to add a barrier method • Note: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period and for 28 days after study drug discontinuation.
* Evidence of clinically significant disease (e.g., cardiovascular, respiratory, gastrointestinal, renal, or infectious disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Any medical or other condition that in the opinion of the investigator(s) would preclude the participant's participation in a clinical study
* Active and current use of illegal recreational drugs
* Currently enrolled in another interventional clinical study or used any investigational drug or device within the past 28 days preceding informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Texas Oncology, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Hutson TE, Michaelson MD, Kuzel TM, Agarwal N, Molina AM, Hsieh JJ, Vaishampayan UN, Xie R, Bapat U, Ye W, Jain RK, Fishman MN. A Single-arm, Multicenter, Phase 2 Study of Lenvatinib Plus Everolimus in Patients with Advanced Non-Clear Cell Renal Cell Carcinoma. Eur Urol. 2021 Aug;80(2):162-170. doi: 10.1016/j.eururo.2021.03.015. Epub 2021 Apr 16. PMID 33867192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in the United States from 20 February 2017 to 2 November 2021.
Pre-assignment Details: A total of 41 participants were enrolled (signed inform consent form) and screened, of which 10 were screen failures and 31 participants received the study treatment.
Groups:
- Lenvatinib 18 mg/Day + Everolimus 5 mg/Day: Participants received initial dose of lenvatinib 18 milligrams per day (mg/day) (one 10-milligram [mg] capsule and two 4-mg capsules), orally once daily and initial dose of everolimus 5 mg/day (5-mg tablets), orally once daily in immediate succession approximately at the same time each morning (consistently either with or without food) in 28-day (4-week) cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or discontinuation by sponsor. Lenvatinib dose reduction was permitted from 18 mg/day to 14, 10, and 8 mg/day, and everolimus dose reduction was permitted from 5 mg/day to 5 mg every other day to manage toxicity, when required.
Period: Overall Study
Arm/Group | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day
Started | 31
Completed | 7
Not Completed | 24
Not completed — Death | 21
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included participants who received at least 1 dose of the study drugs.
Groups:
- Lenvatinib 18 mg/Day + Everolimus 5 mg/Day: Participants received initial dose of lenvatinib 18 mg/day (one 10-mg capsule and two 4-mg capsules), orally once daily and initial dose of everolimus 5 mg/day (5-mg tablets), orally once daily in immediate succession approximately at the same time each morning (consistently either with or without food) in 28-day (4-week) cycles until disease progression, development of unacceptable toxicity, withdrawal of consent, or discontinuation by sponsor. Lenvatinib dose reduction was permitted from 18 mg/day to 14, 10, and 8 mg/day, and everolimus dose reduction was permitted from 5 mg/day to 5 mg every other day to manage toxicity, when required.
Arm/Group | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. ORR was defined as the percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first dose of study drug to the date of the first documentation of disease progression or death, whichever occurred first (up to approximately 3 years 9 months)
Population: The FAS included participants who received at least 1 dose of the study drugs.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day
Number analyzed (Participants) | 31
percentage of participants | 25.8 [11.9 to 44.6]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was assessed by investigator per RECIST v1.1, defined as time from date of first dose of study drug to date of first documentation of progressive disease (PD) or death whichever occurred first. PD: greater than or equal to (>=) 20% increase in sum of diameters of target lesions, reference-smallest sum recorded in study (sum at baseline if that was smallest). Sum of diameters must have absolute increase of >=5 mm. Appearance of >=1 new lesions also considered PD. PFS was analyzed using Kaplan Meier method. PFS was censored on date of last adequate radiologic assessment prior to new anticancer therapy, more than one missed visits, treatment discontinuation, and cutoff date when no PD or death occurred before any of these (on first dose of study treatment if no adequate post baseline tumor assessment was available), per publication by Food and Drug Administration (FDA) 'Guidance for Industry Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics (2007).
Time Frame: as for outcome 1
Population: The FAS included participants who received at least 1 dose of the study drugs.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day
Number analyzed (Participants) | 31
months | 13.11 [5.49 to 24.21]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study drug until the date of death from any cause. OS was analyzed using Kaplan Meier method. In the absence of death before data cutoff, participants were censored either at the date last known to be alive or the date of data cutoff, whichever came earlier. Participants were followed for survival every 12 weeks after the end of treatment visit. If a clinic visit was not feasible, follow-up information was obtained via telephone or email.
Time Frame: From the date of the first dose of study drug until the date of death from any cause (up to approximately 4 years 8 months)
Population: The FAS included participants who received at least 1 dose of the study drugs.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day
Number analyzed (Participants) | 31
months | 16.33 [9.23 to 33.22]

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse events are reported from the first dose of study drug up to 28 days following last dose of study drug, or until resolution of adverse event, whichever occurred first (up to approximately 3 years 10 months) and as planned All-cause mortality is reported from the date of the first dose of study drug until the date of death from any cause (up to approximately 4 years 8 months)
Arm/Group | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day
All-Cause Mortality (participants affected / at risk) | 21/31
Serious Adverse Events (participants affected / at risk) | 12/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day (N=31)
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
International normalised ratio increased (Investigations) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Sepsis (Infections and infestations) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 18 mg/Day + Everolimus 5 mg/Day (N=31)
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cyanosis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Stress cardiomyopathy (Cardiac disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 6
Dry eye (Eye disorders) | 1
Eye swelling (Eye disorders) | 3
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 4
Anal fissure (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 18
Odynophagia (Gastrointestinal disorders) | 1
Oral dysaesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 4
Retching (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 12
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 1
Chills (General disorders) | 2
Crepitations (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 22
Influenza like illness (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 3
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 2
Furuncle (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Respiratory syncytial virus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 4
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Accidental overdose (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Rib fracture (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 1
Aspartate aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 3
Blood creatinine increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 3
Blood urea increased (Investigations) | 1
Heart sounds abnormal (Investigations) | 1
Lipase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
Platelet count increased (Investigations) | 1
Specific gravity urine increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 4
Fluid retention (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dizziness postural (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Hepatic encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Irregular sleep wake rhythm disorder (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Radicular pain (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Ulnar nerve palsy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 7
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 3
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 9
Renal pain (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Sensitive skin (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 4
Jugular vein thrombosis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Asymptomatic bacteriuria (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Injection site abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Lipids increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT02915783/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT02915783/SAP_001.pdf